CLINICAL TRIAL: NCT02440516
Title: Standardized Comprehensive Two-month Ambulatory Neurorehabilitation Program for Patients With Multiple Sclerosis: a Randomized-controlled Trial
Brief Title: Standardized Ambulatory Neurorehabilitation Program for Patients With Multiple Sclerosis
Acronym: "MS-Fit"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015_04_29
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
Keywords: Standardized; Physical therapy; occupational therapy; quality of life; disability; activities of daily living; ambulatory therapy; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurorehabilitation program (Active Comparator): Standardized comprehensive ambulatory neurorehabilitation program
  Interventions: Other: Early treatment group
- Waiting list (Placebo Comparator): Waiting list
  Interventions: Other: Late treatment group

INTERVENTIONS:
Other: Early treatment group — Physical- and occupational Therapy
  Arms: Neurorehabilitation program
Other: Late treatment group — Waiting list - then Physical- and occupational Therapy
  Arms: Waiting list

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) and the most common cause of non-traumatic disability in young adults in western countries. Despite increasing therapeutic options to ameliorate the disease course, most patients suffer from persistent neurological deficits over time.

Disability in MS has a negative impact on patients life's impairing activities of daily living (ADL) and quality of life (QoL) and leading to loss of work and the need providing care. This results in tremendous socioeconomic burden.

Disease-modifying treatments prevent disability progression in variable extent. However no drugs are available ameliorate persistent disability in MS. Therefore, exercise training as well as physical and occupational therapies are important in the symptomatic treatment of MS.

Physical and occupational therapy is usually performed close to patients home by therapist with different professional background in a non-standardized way.

The investigators therefore aim to develop a standardized comprehensive ambulatory neurorehabilitation program, integrating task oriented circuit training for MS patients to improve disability, ADL and QoL that can be easily adopted in other ambulatory or hospital settings.

DETAILED DESCRIPTION:
Background

Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) and the most common cause of non-traumatic disability in young adults in western countries. The incidence of MS is low in childhood and increases after the age of 18, reaching a peak between 20 and 40 years (mean age of 30 years) with women being affected approximately 2-5 years earlier than men. In Switzerland the incidence is thought to be 4:100.000 with approximately 12.500 affected patients.

Despite increasing therapeutic options to ameliorate the disease course, most patients suffer from persistent neurological deficits over time.

Neurologic symptoms can be manifold and are highly variable amongst patients. They include loss of vision, sensorimotor defects, impaired manual dexterity, ataxia, apraxia, gait disturbances, bladder- and bowl problems, fatigue, cognitive dysfunctions and others, which alone, or in combination, lead to disability in MS patients. Disability in MS has a negative impact on patients life's impairing activities of daily living (ADL) and quality of life (QoL) and leading to loss of work and the need providing care. This results in tremendous socioeconomic burden.

Disease-modifying treatments prevent disability progression in variable extent. However no drugs are available ameliorate persistent disability in MS. Therefore, exercise training as well as physical and occupational therapies are important in the symptomatic treatment of MS. Intensive task oriented circuit training has been shown to be effective in stroke improving gait, and several ADL. Some pilot randomized controlled trials in MS demonstrated exercise training being able to improve muscular strength, aerobic capacity and ambulatory performance as well as fatigue, balance and gait. Furthermore, specific therapies improve manual dexterity, coordination and mobilization in MS patients as well. Although, so far no randomized trial has been done to prove the effectiveness of task oriented circuit training in MS.

Physical and occupational therapy is usually performed close to patients home by therapist with different professional background in a non-standardized way.

The investigators therefore aim to develop a standardized comprehensive ambulatory neurorehabilitation program, integrating task oriented circuit training for MS patients to improve disability, ADL and QoL that can be easily adopted in other ambulatory or hospital settings.

Objective

To evaluate the impact of a standardized comprehensive ambulatory neurorehabilitation program on disability in patients with multiple sclerosis measured by performance based test of the upper and lower extremities and by patient recorded outcome measures regarding functioning of the upper and lower extremities, activities of daily living and quality of life.

The investigators hypothesize that this training program will improve disability, activities of daily living and quality of live in MS patients.

Methods

Prospective double center, randomized, cross-over study. Consecutive MS patients that complain about disability that affects ADL and/or QoL will be recruited to participate in a comprehensive ambulatory neurorehabilitation program. Afterwards baseline measurements will be performed and patients will be randomized 1:1 into the early treatment group or the delayed treatment group in groups of four using sealed envelopes. The early treatment group starts the neurorehabilitation program whereas in the delayed treatment group, patients will be put on a waiting list for two months. After two months, outcome measurements will be collected. Patients of the early treatment group stop the neurorehabilitation program and patients of the delayed treatment group start the neurorehabilitation program for two months ("cross-over design"). Two months after ending the program, each group will be retested.

ELIGIBILITY:
Inclusion Criteria:

* MS patients with relapsing-remitting MS (RRMS), secondary-progressive MS (SPMS) or primary progressive MS (PPMS)
* Age between 18 and 75 years
* Written informed consent
* Patient complains about MS related disability that affects ADL and/or QoL

Exclusion Criteria:

* A relapse that started within 60 days prior to screening
* Rapidly progressive disease
* Any disease/condition that causes neurological deficits or disability besides MS
* A history of drug abuse in the 12 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Multiple Sclerosis Impact Scale 29 (MSIS-29) | 2 - 4 months
  The Multiple Sclerosis Impact Scale (MSIS-29) is valid and reliable (ICC 0.80 - 0.87) in measuring the impact of MS on ADL.It contains 29 items comprising to a physical (MSIS-29 physical) and psychological impact scale (MSIS-29 psychological). All items are scored from 'not at all' to 'extremely' on a five-point Likert scale.

SECONDARY OUTCOMES:
Change from baseline in Coin Rotation Task (Heldner et al. 2014) | 0 - 2 - 4 months
  The Coin Rotation Task (CRT) has been validated in assessing manual dexterity in patients with MS. Patients had to rotate a 50 Swiss Rappen coin (corresponding to a dime or 2-cent Euro coin) as fast as possible between their thumb, index and middle finger. The time to perform 20 half turns was measured twice on both hands and mean values were taken for each hand. If patients could not perform the CRT due to impaired manual dexterity, an arbitrarily chosen value of 300 seconds was taken.
Change from baseline in Timed Up and Go (TUG) (Nilsagard et al. 2007) | 0 - 2 - 4 months
  The Timed Up and Go test (TUG) is a test used to assess a person's mobility. It uses the time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down.
Change from baseline in Nine-hole-Peg Test (NHPT) (Gookin et al. 1988) | 0 - 2 - 4 months
  The Nine Hole Peg Test (9HPT) is reliable (ICC values 0.80-0.99), valid and sensitive in detecting impaired dexterity in patients with MS. Patients were seated at a table with a shallow container holding nine pegs and a plastic block with nine empty holes. All pegs had to be put one at a time into the holes and then removed again one at a time into the shallow container. The time to complete the task was recorded twice on both hands and mean values were taken for each hand. If patients could not perform the CRT due to impaired manual dexterity, an arbitrarily chosen value of 300 seconds was taken.
Change from baseline in 25-Foot Walk Test (25-FWT) (Cohen et al. 2014) | 0 - 2 - 4 months
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the MSFC to be administered at each visit. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Change from baseline in EDSS | 0 - 2 - 4 months
Change from baseline in Rand 36 | 0 - 2 - 4 months
  The RAND-36 is a license free version of the Short-Form Health Survey-36 (SF-36) containing eight scales.15 Each scale comprises two to ten items, and makes up to two summary measures. The scales measuring "physical functioning", "role-physical", "bodily pain" and "general health" form the "physical health summary score". The scales measuring "vitality", "social functioning", "role-emotional" and "mental health" form the "mental health summary score".
Change from baseline in Fatigue Severity Scale | 0 - 2 - 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Kamm, MD, Principal Investigator — Department of Neurology, Cantonal hospital Luzern
Locations (2):
- Switzerland (2):
  - Department of Neurology, Bern University Hospital, Bern
  - Department of Neurology, Cantonal hospital Luzern, Lucerne

REFERENCES:
- [Background] Kamm CP, Uitdehaag BM, Polman CH. Multiple sclerosis: current knowledge and future outlook. Eur Neurol. 2014;72(3-4):132-41. doi: 10.1159/000360528. Epub 2014 Jul 30. PMID 25095894
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. How responsive is the Multiple Sclerosis Impact Scale (MSIS-29)? A comparison with some other self report scales. J Neurol Neurosurg Psychiatry. 2005 Nov;76(11):1539-43. doi: 10.1136/jnnp.2005.064584. PMID 16227547
- [Result] Motl RW, Pilutti LA. The benefits of exercise training in multiple sclerosis. Nat Rev Neurol. 2012 Sep;8(9):487-97. doi: 10.1038/nrneurol.2012.136. Epub 2012 Jul 24. PMID 22825702
- [Derived] Lehmann I, Thaler I, Luder G, Damm U, Walti C, Steinheimer S, Verra ML, Muri RM, Nyffeler T, Vanbellingen T, Kamm CP. Standardized, comprehensive, hospital-based circuit training in people with multiple sclerosis: results on feasibility, adherence and satisfaction of the training intervention. Eur J Phys Rehabil Med. 2020 Jun;56(3):279-285. doi: 10.23736/S1973-9087.20.06191-2. Epub 2020 Mar 30. PMID 32225136